CLINICAL TRIAL: NCT01945047
Title: Phase 2 Optimization of the Antidepressant Action of Ketamine in Treatment-Resistant Depression and Investigations on Its Mechanism of Action
Brief Title: Action of Ketamine in Treatment-Resistant Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Pierre Blier, Endowed Chair and Director of Mood Disorders Research Unit, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: REB2012023
Record Dates: First submitted 2013-05-22; First posted 2013-09-18 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Treatment-resistant Depression
Keywords: depression; treatment; ketamine; ottawa; treatment-resistant; infusion
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): During Phase 1 patients will be randomly assigned to receive ketamine or active placebo.
  Interventions: Drug: Ketamine
- Midazolam (Active Comparator): In phase 1 patients will be randomized to receive active placebo
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — Intravenous Bolus infusion Ketamine Hydrochloride 0.50 mg/mL over 40 minutes
  Other Names: Ketamine Hydrochloride; Kevlar
  Arms: Ketamine
Drug: Midazolam — Bolus infusion of Midazolam Hydrochloride 1 mg/mL over 40 minutes
  Other Names: Midazolam Hydrochloride; Midazolam HCL
  Arms: Midazolam

SUMMARY:
Depression carries the largest burden of all medical disorders in middle to high income countries, as determined by the World Health Organization. Despite many antidepressant strategies, only a third of patients get well after their first treatment and a third remain ill after several treatments. Moreover, antidepressant treatments all have a delayed action ranging up to several weeks.

Ketamine (KET) has been used for decades as a sedative and anesthetic. In treatment-resistant depressed patients(TRD), an intravenous dose much lower than necessary for anesthesia may produce a robust antidepressant effect and may even abolish suicidal thoughts within hours, peaking within 24 hours. But, its antidepressant effect generally lasts only days.Previous studies examining KET in TRD have been critiqued for lack of an effective placebo measure due to brief perceptual experiences associated with KET. Thus, the current study compares KET against a short-acting sedative. The phases of this study compare response to a single KET injection to 6 injections over 2 weeks. Next, KET responders are given 1 injection a week for 3 weeks of either KET or the sedative agent to determine if beneficial effects of KET are maintained, and to assess duration of its benefits after repeated administration. The genetic profile of patients for a substance promoting contacts between cells and brain will be determined to investigate if response to KET could be predicted with that blood test. This substance, as well as several chemicals that produce inflammation, will also be measured in the blood to investigate their role in the effect of KET. Patients will receive, in total, no more than the equivalent of two to three anesthetic dose of KET. Results from this study will help establish the beneficial effects of a single KET injection as a rapid intervention for major depression, and to investigate the possibility of obtaining a prolonged antidepressant effect with repeated injections.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) carries worldwide the largest burden of diseases among mental, neurological, and substance-use disorders measured in Disability Adjusted Life Years (DALYs), according to the World Health Organization (WHO).1 In turn, MDD has the highest DALYs in middle to high income countries, with ischemic cardiac diseases being second.2 Although there are effective treatments for MDD, a large proportion of patients do not achieve remission even after several attempts, and any significant response, when it manifests itself, takes place a delay of a few weeks.3,4 There is always urgency to treat MDD because although patients may have been ill for several weeks, months, and sometimes years, they are often in a crisis situation when they consult. The nature of the crisis may be familial, financial/professional, or the consultation may take place because of intense personal suffering, possibly involving suicidal ideation. Consequently, rapid therapeutic action and high remission rates represent the two major unmet needs for MDD.

In the last few years, considerable attention has been dedicated to the glutamate system as a possible contributor of the antidepressant response. The most striking breakthrough has been the rapid antidepressant response of intravenous ketamine using doses that are about a quarter of the routinely utilized anesthetic dose in children and adults.5,6 Unlike many anesthetic agents, ketamine does not depress cardiovascular and respiratory parameters.7 The primary action of ketamine is to block N-Methyl-D-Aspartate (NMDA) receptors. The antidepressant response to ketamine often manifests itself within a few hours, but is generally maximal after 24 hours.8 Importantly, a single infusion produces in the most subjects a robust decrease of suicidal ideation.9,10 The drawback of this approach is, however, that its benefits generally disappear within a week.6 Consequently, much clinical work remains to be carried out in order to better understand and maintain the antidepressant response of ketamine.

Specific aim #1: The first aim of this proposal is to characterize the antidepressant action of a single dose of ketamine in a truly double-blind paradigm. Indeed, even the low doses of ketamine (0.2-0.5 mg/kg)8,11 produce mild derealization and therefore the use a mere saline solution in prior studies has been inadequate as a control.

1. To show that the infusion of a low dose of the short-acting benzodiazepine midazolam will serve as an adequate active control for ketamine. It is hypothesized that because midazolam produces marked sedation, it will serve as an adequate control.
2. To determine if the brain-derived neutrophic factor (BDNF) mediates the antidepressant response. In mice, a VAL/MET polymorphism for the BDNF gene, ketamine is devoid of effects. The influence of this polymorphism will be evaluated in patients.

Specific aim #2: The second goal of this proposal is to attempt enhancing and prolonging the antidepressant effect of ketamine by giving it repeatedly at a rate of three infusions per week for two consecutive weeks.

1. To assess whether ketamine responders will improve further after a six infusions over two weeks. It is hypothesized that ketamine non-responders following a single infusion will not show a significant improvement with repeated infusions of ketamine at a dose of 0.5 mg/kg given three times a week for two weeks, but that in responders repeated ketamine will produce a more robust and sustained antidepressant action than a single infusion.
2. To assess whether the inflammatory status of the depressed patients is altered by the response to ketamine. Pro-inflammatory mediators and cortisol are generally elevated in depression while melatonin is decreased. These anomalies are typically restored with effective treatments. This will be investigated in the light of the rapid antidepressant effect of ketamine.

Specific aim #3: The third goal of this proposal is to prolong the antidepressant effect of ketamine. In this third consecutive phase of the project, ketamine-responsive patients will receive ketamine on a once weekly basis.

1)To demonstrate that the antidepressant effect of ketamine will be sustained over four weeks using a single infusion per week. The antidepressant response to a single infusion of ketamine disappears within 7 days. It is hypothesized that repeated infusions of ketamine, at an interval of one week for four weeks, will maintain the antidepressant effect.

2)To assess how long the antidepressant effect of repeated ketamine infusions will last in follow up. After the first three phases of this project that will last about eight weeks, the average duration of a standard antidepressant medication trial, the responders will be monitored to follow their clinical evolution. It is hypothesized that the responders will show a longer maintenance of their response than after the first infusion in phase one of the project.

1. Phase I: the double-blind crossover. After patients will have been deemed eligible to participate in the study, blood will be drawn for genotyping and various assays (BDNF Val/Met, BDNF, morning melatonin and salivary cortisol, C-reactive protein, IL-1β, IL-2, IL-6, IL-8, IL-12, IFN-γ, TNF-α, and anti-inflammatory factors IL-4 and IL-10, as previously done in our laboratory).101-102 They will be randomized to receive intravenously either 0.5 mg/kg of ketamine (the readily available racemic mixture) or 30 µg/kg of midazolam as a 250 ml infusion (prepared in our unit) over 40 minutes, given by a research nurse in the presence of a study physician. Their antidepressant drug regimen will not be altered throughout the study. A clinician will evaluate their clinical status prior to the infusion, using the Montgomery-Asberg Depression Rating Scale (MADRS)103 and the Clinical Global Intensity-Severity (CGI-S)104 and the patients will rate themselves using the Quick Inventory Depressive Symptoms-Self-report (QIDS-SR)105 and a self-report questionnaire rating suicidality. The patients will be assessed using the Brief Psychiatric Rating Scale-positive symptom scale106 at baseline (before the infusion), time 0 (immediately after infusion is complete), then at 60 and 120 minutes post time 0. The CGI-Improvement (CGI-I)104 will be used to obtain a clinical evaluation of overall change of their condition after two hours before discharging the patients two hours after the infusion. The patients will come in the next day for an evaluation using the MADRS, CGIs, and the QIDS-SR and will be asked to guess what drug they received. Four days after the infusion, the patients will repeat the QIDS-SR at home, and they will come in for an evaluation at day 7. If the patients did not respond, or if they returned to 80% of their MADRS score before the infusion, they will receive either ketamine or midazolam to complete the crossover protocol. If the patients are maintaining more than a 20% improvement of their baseline MADRS score, they will be asked to come in on a weekly basis for an assessment, and will be asked to complete a QIDS-SR twice a week (at days 10, 14, 18, 21, and so on) in order to assess how long the therapeutic effect lasts. Patients who have not response to their second infusion or those found to have relapsed during the weekly follow-up visits, will continue into phase II. Patients who are unable, ineligible, or unwilling to enter phase II will be given a recommended treatment plan and returned to their family physician with a consultation plan, or additional/alternative treatment options at the discretion of the study physician.

   In order to obtain an objective measure of their activity level and of the pattern of their sleep-wake cycle, patients will wear an actimeter watch for several days during screening and throughout the protocol. The data will be downloaded weekly during the visits.
2. Phase II: the repeated treatment over two weeks. Once patients are deemed not to have responded to the second infusion or have lost their improvement (relapsing to a MADRS score over 80% of their baseline score prior to the second infusion), they will receive repeated ketamine infusions (0.5 mg/kg). They will be given 3 infusions per week for two weeks. On visit 6 of phase 2 the patients will be assessed using the Brief Psychiatric Rating Scale-positive symptom scale106 at baseline (before the infusion), time 0 (immediately after infusion is complete), then at 60 and 120 minutes post time 0. Their clinical status will be assessed prior to each infusion using the MADRS, the CGI-S, the CGI-I, and they will rate themselves using the QIDS-SR and a self-report questionnaire rating suicidality. Patients will be assessed two to three days after the sixth infusion. The ratings throughout phase II will help determine whether repeated administration produces a greater and sustained improvement than a single infusion. Biological assays will be repeated at the end of Phase II.
3. Phase III: the repeated treatment over four weeks and the naturalistic follow-up.

Two to three days after the sixth infusion, patients not achieving a 50% improvement of their MADRS score, when compared to their baseline score prior to the first of the six infusions, will be taken out of the study and offered to be treated in our Research Unit using additional pharmacological and/or psychotherapeutic approaches. Patients improving by 50% or more on the MADRS scale will receive ketamine once a week for four weeks. They will be assessed using the same scales as mentioned above prior to each infusion. Patients will be assessed two to three days after the fourth weekly infusion. The ratings throughout phase III will help determine whether repeated administration of ketamine is effective to maintain the beneficial action of a relatively more intense regimen of ketamine.

Monitoring of the patients reaching more than 80% or more of their MADRS score, when compared to their baseline score prior to the last four infusions, will cease and will be offered to be treated in our Research Unit using additional pharmacological and/or psychotherapeutic approaches. Patients maintaining more than 20% improvement will be assessed weekly to determine how long the therapeutic effects of ketamine last. Biological assays will be repeated at the end of Phase III.

ELIGIBILITY:
Inclusion Criteria:

* Only participants from the Ottawa area will be considered
* Provision of written informed consent before initiation of any study- related procedures.
* Documented primary Axis I clinical diagnosis meeting criteria from the DSM-IV13 for MDD, as confirmed by the MINI.98
* Failure to respond adequately to at least two antidepressant medication trials and two augmentation strategies. One augmentation strategy may include a noradrenergic dose of venlafaxine (225 mg/day) or duloxetine (120 mg/day), given their dual mechanism of action99,100 and a 12-week cognitive behavioural or interpersonal therapy
* MADRS total score of ≥ 25 at screening and randomization, with no more than 20% improvement between these two visits.
* Female subjects of childbearing potential must have a negative urine pregnancy test at enrolment (Visit 1) and be willing to use a reliable method of birth control (i.e., double-barrier method, oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, intrauterine device, or tubal ligation) during the study.
* Abstain from consuming grapefruit juice (a potent 3A4 cytochrome inhibitor) on the day of the infusions as it may slow down the elimination of midazolam and possibly ketamine.
* Be able to understand and comply with the requirements of the study, as judged by the investigator(s).

Exclusion Criteria:

* Subjects with a diagnosis of DSM-IV Axis II disorder which has a major impact on the subject's current psychiatric status.
* Depression secondary to stroke, cancer or other severe medical illnesses.
* Prior or current substance or alcohol abuse or dependence (except for caffeine or nicotine dependence), as defined in DSM-IV criteria.
* A positive drug screen.
* Unwilling to maintain their current antidepressant regimen. infusions.
* Unwilling or able to hold benzodiazepines on the day prior and that of the Unwilling to discontinue any narcotic for a minimum of 5 drug half-lives prior to infusions.
* Pregnant or lactating, or is of childbearing potential and not willing to use an approved method of contraception during the study.
* Evidence of clinically relevant disease, e.g., renal or hepatic impairment, significant coronary artery disease (myocardial infarct within a year prior to initial randomization), cerebrovascular disease, viral hepatitis B or C, acquired immunodeficiency syndrome.
* A clinical finding that is unstable or that, in the opinion of the investigator(s), would be negatively affected by the study medication or that would affect the study medication (e.g., diabetes mellitus, hypertension, unstable angina).
* Liver function tests AST and ALT three times the upper normal limit at screening.
* Uncorrected hypothyroidism or hyperthyroidism. Subjects needing a thyroid hormone supplement to treat hypothyroidism must have been on a stable dose of the medication for 30 days prior to enrolment (Visit 1).
* Clinically significant deviation from the reference range in clinical laboratory test results as judged by the investigator(s).
* ECG results considered clinically significant as determined by the investigator(s).
* History of seizure disorder, except febrile convulsions.
* Subjects who in the investigator(s) opinion will require psychotherapy (other than supportive psychotherapy) during the study period, unless psychotherapy has been ongoing for a minimum of 2 months prior to Visit 2.
* Known history of intolerance or hypersensitivity to ketamine or midazolam.
* Any other condition that, in the opinion of the investigator(s) would adversely affect the subject's

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of Ketamine over Midazolam in double blind study for efficacy of relief for Major Depressive Disorder | 2 weeks
  Phase 1 double blind treatment with Ketamine or Midazolam then crossover. Will assess efficacy of each for relief of Major Depressive Symptoms through assessment using the HAMD17.

SECONDARY OUTCOMES:
Ketamine for use in relief of Major Depressive Disorder over repeated administration | 6 weeks
  Repeated infusion of ketamine in phases 2 and 3 to determine efficacy over extended treatment period.We will assess effectiveness for treatment of depression by administering the Montgomery-Asberg Depression Rating Scale (MADRS)to assess severity of depressive symptoms. MADRS will be given before and after each infusion and at follow up visits to monitor changes.
To determine the role of genetic polymorphisms in the participants response to ketamine infusion | 2 weeks
  Patients will be genotyped for a VAL/MET polymorphism for the brain-derived neutrophic factor (BDNF)gene to see whether presence or absence of the polymorphism mediates their antidepressant response.

OTHER OUTCOMES:
Cortisol, melatonin, and inflammatory mediators will be assessed to examine changes occurring during treatment with ketamine | 8 weeks
  Pro-inflammatory mediators and cortisol are generally elevated in depression while melatonin is decreased. These anomalies are typically restored with effective treatments. This will be investigated in the light of the rapid antidepressant effect of ketamine.
  During phase 1, patients will provide samples of saliva for morning melatonin and salivary cortisol at 1)Randomization, 2)Phase 2,infusion 6, 3)Phase 3, infusion 4. Collected for 2 days: Immediately upon waking;30 minutes later;1 hour later;Mid-day.
  Inflammatory mediators will be assessed to determine changes occurring throughout treatment. Two blood samples will be drawn at each of the following study visits: Randomization;Phase 2, infusion 6;Phase 3, infusion 4 We will examine C-reactive protein, IL-1β, IL-2, IL-6, IL-8, IL-12, IFN-γ, TNF-α, and anti-inflammatory factors IL-4 and IL-10.
Effects of ketamine infusion compared to midazolam | 2 weeks
  A clinician will evaluate their clinical status prior to the infusion, using the Montgomery-Asberg Depression Rating Scale (MADRS) and the Clinical Global Intensity-Severity (CGI-S) and the patients will rate themselves using the Quick Inventory Depressive Symptoms-Self-report (QIDS-SR)105 and a self-report questionnaire rating suicidality. The patients will be assessed using the Brief Psychiatric Rating Scale-positive symptom scale at baseline (before the infusion), time 0 (immediately after infusion is complete), then at 60 and 120 minutes post time 0. The CGI-Improvement (CGI-I) will be used to obtain a clinical evaluation of overall change of their condition after two hours before discharging the patients two hours after the infusion. We will compare the scores on the scales used in ketamine infusion verses midazolam to evaluate whether ketamine is superior but also whether midazolam is an effective control (patients feel some effects similar to ketamine infusion)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Blier, M.D, Ph.D, Principal Investigator — University of Ottawa
Locations (1):
- Institute of Mental Health Research, Royal Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Phillips JL, Van Geel A, Burhunduli P, Vasudev D, Batten LA, Norris S, Talbot J, Ortiz A, Owoeye O, Blier P. Assessment of Objective and Subjective Cognitive Function in Patients With Treatment-Resistant Depression Undergoing Repeated Ketamine Infusions. Int J Neuropsychopharmacol. 2022 Dec 12;25(12):992-1002. doi: 10.1093/ijnp/pyac045. PMID 35931041
- [Derived] de la Salle S, Phillips JL, Blier P, Knott V. Electrophysiological correlates and predictors of the antidepressant response to repeated ketamine infusions in treatment-resistant depression. Prog Neuropsychopharmacol Biol Psychiatry. 2022 Apr 20;115:110507. doi: 10.1016/j.pnpbp.2021.110507. Epub 2021 Dec 28. PMID 34971723
- [Derived] Phillips JL, Norris S, Talbot J, Birmingham M, Hatchard T, Ortiz A, Owoeye O, Batten LA, Blier P. Single, Repeated, and Maintenance Ketamine Infusions for Treatment-Resistant Depression: A Randomized Controlled Trial. Am J Psychiatry. 2019 May 1;176(5):401-409. doi: 10.1176/appi.ajp.2018.18070834. Epub 2019 Mar 29. PMID 30922101